CLINICAL TRIAL: NCT04904549
Title: A Parallel-group, Phase III, Multi-stage, Modified Double-blind, Multi-armed Study to Assess the Efficacy, Safety, and Immunogenicity of Two SARS-CoV-2 Adjuvanted Recombinant Protein Vaccines (Monovalent and Bivalent) for Prevention Against COVID-19 in Adults 18 Years of Age and Older as a Primary Series and Open-label Extension to Assess Immunogenicity, Safety, Efficacy of a Monovalent Booster Dose of SARS-CoV2 Adjuvanted Recombinant Protein Vaccine
Brief Title: Study of Monovalent and Bivalent Recombinant Protein Vaccines Against COVID-19 in Adults 18 Years of Age and Older
Acronym: VAT00008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAT00008; U1111-1264-3238 (Registry Identifier: ICTRP); VAT00008 (Other: Sanofi Identifier)
Record Dates: First submitted 2021-05-26; First posted 2021-05-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study is designed to demonstrate clinical efficacy of each of the two SARS-CoV-2 adjuvanted recombinant protein vaccines (monovalent and bivalent). In Stage 1, the monovalent vaccine will be evaluated against a placebo control. In Stage 2, the bivalent vaccine will be assessed against a placebo control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For initial, double-blind, primary series design of study: participants, outcome assessors, Investigators, laboratory personnel, and sponsor trial staff are blinded to intervention group; and those preparing the study interventions are unblinded to vaccine assignment group.
  For crossover / booster design of study (Stage 1 and Stage 2): unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1: SARS-CoV-2 vaccine (Experimental): 2 injections of monovalent SARS-CoV-2 vaccine at Day 1 and Day 22
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (monovalent D614) (primary series); Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (monovalent B.1.351) (booster dose) >= 4 months after last vaccination
- Stage 1: Placebo (Placebo Comparator): 2 injections of placebo at Day 1 and Day 22
  Interventions: Biological: Placebo; Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent D614)(primary series)& SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent B.1.351)(booster dose)>=4 months after last vaccination
- Stage 2: SARS-CoV-2 vaccine (Experimental): 2 injections of bivalent SARS-CoV-2 vaccine at Day 1 and Day 22
  Interventions: Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (bivalent D614 + B.1.351) (primary series); Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (monovalent B.1.351) (booster dose) >= 4 months after last vaccination
- Stage 2: Placebo (Placebo Comparator): 2 injections of placebo at Day 1 and Day 22
  Interventions: Biological: Placebo; Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent D614)(primary series)& SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent B.1.351)(booster dose)>=4 months after last vaccination

INTERVENTIONS:
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (monovalent D614) (primary series) — Pharmaceutical form: emulsion for injection. Route of administration: intramuscular injection
  Arms: Stage 1: SARS-CoV-2 vaccine
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (bivalent D614 + B.1.351) (primary series) — Pharmaceutical form: emulsion for injection. Route of administration: intramuscular injection.
  Arms: Stage 2: SARS-CoV-2 vaccine
Biological: Placebo — Pharmaceutical form: liquid. Route of administration: intramuscular administration.
  Arms: Stage 1: Placebo; Stage 2: Placebo
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine (monovalent B.1.351) (booster dose) >= 4 months after last vaccination — Pharmaceutical form: emulsion for injection. Route of administration: intramuscular injection.
  Arms: Stage 1: SARS-CoV-2 vaccine; Stage 2: SARS-CoV-2 vaccine
Biological: SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent D614)(primary series)& SARS-CoV-2 adjuvanted recombinant protein vaccine(monovalent B.1.351)(booster dose)>=4 months after last vaccination — Pharmaceutical form: emulsion for injection. Route of administration: intramuscular injection.
  Arms: Stage 1: Placebo; Stage 2: Placebo

SUMMARY:
The purpose of this Phase III study is to assess the efficacy, safety, and immunogenicity of two CoV2 preS dTM-AS03 vaccines (monovalent and bivalent) as part of primary series vaccinations in a multi-stage approach, as well as a booster injection of a CoV2 preS dTM-AS03 vaccine, in adults 18 years of age and older.

A total of approximately 21 046 participants are planned to be enrolled (5080 per study intervention group in Stage 1 and 5443 per study intervention group in Stage 2).

Initial, double-blind, primary series study design is planned for 365 days post-last Initial injection (ie, approximately 386 days total) for each participant.

Based on decisions of the Study Oversight Group, Stage 1 and Stage 2 participants will be invited to participate in an unblinded Crossover / Booster study design with duration as follows:

* For participants who initially received vaccine: 12 months post-booster (ie, approximately 18 to 24 months)
* For participants who initially received placebo: ≥ 4 months post-last dose of the primary series + 12 months post-booster (ie, approximately 28 to 34 months)
* For participants who do not consent to continue in the unblinded Crossover / Booster part of the study, all study procedures will be stopped and participants will be discontinued from the study.

DETAILED DESCRIPTION:
The duration of participation in the initial, double-blind, primary series design of the study will be approximately 365 days post-last injection (ie, approximately 386 days total) for each participant.

Based on decisions of the Study OG, Stage 1 and Stage 2 participants will be invited to participate in an unblinded Crossover / Booster study design with duration as follows:

* For participants who initially received vaccine: 12 months post-booster (ie, approximately 18 to 24 months)
* For participants who initially received placebo: ≥ 4 months post-last dose of the primary series + 12 months post-booster (ie, approximately 28 to 34 months)
* For participants who do not consent to continue in the unblinded Crossover / Booster part of the study, all study procedures will be stopped and participants will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on the day of inclusion.
* For persons living with human immunodeficiency virus (HIV), stable HIV infection determined by participant currently on antiretrovirals with CD4 count > 200/mm3.
* SARS-CoV-2 rapid serodiagnostic test performed at the time of enrollment to detect presence of SARS-CoV-2 antibodies.
* Does not intend to receive an authorized/approved COVID-19 vaccine despite encouragement by the Investigator to receive the authorized vaccine available to them at the time of enrollment.
* Informed consent form has been signed and dated
* Able to attend all visits and to comply with all study procedures
* Covered by health insurance, only if required by local, regional or national regulations
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile, or
  * is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first study intervention administration until at least 12 weeks after the second study intervention administration.

A participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 25 hours before any dose of study intervention.

Exclusion Criteria:

* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances.
* Dementia or any other cognitive condition at a stage that could interfere with following the study procedures based on Investigator?s judgment.
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination based on Investigator?s judgment
* Bleeding disorder, or receipt of anticoagulants in the past 21 days preceding inclusion, contraindicating IM vaccination based on Investigator?s judgment.
* Unstable acute or chronic illness that in the opinion of the Investigator or designee poses additional risk as a result of participation or that could interfere with the study procedures.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ? 38.0 C [? 100.4 F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of any vaccine in the 30 days preceding or on the day of the first study vaccination or planned receipt of any vaccine between the first study vaccination and in the 30 days following the second study vaccination except for influenza vaccination, which may be received at any time in relation to study intervention.
* Prior administration of a coronavirus vaccine (SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome).
* Receipt of solid-organ or bone marrow transplants in the past 180 days.
* Receipt of anti-cancer chemotherapy in the last 90 days.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23726 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Occurrences of symptomatic COVID-19 | From ≥ 14 days after the second injection to Day 387
  Symptomatic COVID-19 is defined as virologically-confirmed SARS-CoV-2 infection accompanied by protocol-defined COVID-19-like illness.
Presence of solicited injection site or systemic reactions (collected in the reactogenicity subset) | Within 7 days after vaccination
  Injection site reactions: injection site pain, erythema and swelling. Systemic reactions: fever, headache, malaise, myalgia, arthralgia and chills.
Presence of non-serious unsolicited adverse events (collected in the reactogenicity subset) | Within 21 days after vaccination
  Adverse events other than solicited reactions.
Presence of immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events include unsolicited injection site and systemic adverse events occurring within 30 minutes after injection.
Presence of medically attended adverse events | From Day 1 to Day 387
  Medically attended adverse events will be assessed throughout the study.
Presence of serious adverse events | From Day 1 to Day 387
  Serious adverse events will be assessed throughout the study.
Presence of adverse events of special interest | From Day 1 to Day 387
  Adverse events of special interest will be assessed throughout the study.
Presence of virologically-confirmed SARS-CoV-2 infections and/or symptomatic COVID-19 | From Day 1 to Day 387
  Percentage of participants with positive result for SARSCoV-2 infection by Nucleic Acid Amplification Test (NAAT) on at least one respiratory sample accompanied or not by protocol-defined clinical COVID-19 symptoms.

SECONDARY OUTCOMES:
Occurrences of SARS-CoV-2 infection | From ≥ 14 days after the second injection to Day 387
  SARS-CoV-2 infection is defined as a serologically-confirmed SARS-CoV-2 infection or virologically-confirmed SARS-CoV-2 infection.
Occurrence of severe COVID-19 | From ≥ 14 days after the second injection to Day 387
Occurrences of asymptomatic SARS-CoV-2 infection | From Day 1 to Day 387
  Asymptomatic SARS-CoV-2 infection is defined as SARS-CoV-2 infection, with no reported COVID-19-like illness episodes between enrollment and 14 days after the timepoint at which SARS-CoV-2 infection is ascertained.
Number of days with positive NAAT | From Day 1 to Day 387
Viral copies/mL in respiratory samples | From Day 1 to Day 387
Occurrences of positive NAAT in respiratory samples at each follow-up timepoint during symptomatic COVID-19 | From Day 1 to Day 387
Occurrences of CDC-defined COVID-19 | From Day 1 to Day 387
  Virologically-confirmed SARS-CoV-2 infection with at least one of CDC-defined clinical symptoms.
Occurrences of hospitalized COVID-19 | From Day 1 to Day 387
  Hospitalized COVID-19 is defined as an episode of symptomatic COVID-19 that requires inpatient hospitalization.
Occurrences of symptomatic COVID-19 with severity of moderate COVID-19 or worse. | From Day 1 to Day 387
  Composite endpoint of at least one of moderate or severe COVID-19.
Neutralizing antibody titer | Day 1, Day 22, Day 43, Day 78, Day 134, Day 202, Day 292, and Day 387
Responders, as determined by neutralizing antibody titers | Day 1, Day 22, Day 43, Day 78, Day 134, Day 202, Day 292, and Day 387
  Responders are defined as participants who had baseline values below lower limit of quantification (LLOQ) with quantifiable neutralization titer above assay LLOQ at each pre-defined post-vaccination time point and participants with baseline values above LLOQ with a 4-fold increase in neutralizing antibody
Neutralizing antibody titer fold-rise post-vaccination at all pre-defined time points | Day 1, Day 22, Day 43, Day 78, Day 134, Day 202, Day 292, and Day 387
  Fold-rise in antibody neutralization titer post-vaccination relative to Day 1.
2-fold rise and 4-fold-rise in neutralization antibody titer at all pre-defined time points | Day 1, Day 22, Day 43, Day 78, Day 134, Day 202, Day 292, and Day 387
  Fold-rise in antibody neutralization titer post-vaccination relative to Day 1.
Severity of symptoms associated with symptomatic COVID-19 episode | From Day 1 to Day 387
Occurrences of COVID-19 in each severity rating | From Day 1 to Day 387
  COVID-19 severity score based on the ordinal scale of clinical assessment (7-point ordinal scale)
Death associated with COVID-19 | From Day 1 to day 387

CONTACTS AND LOCATIONS:
Locations (86):
- United States (23):
  - AES - DRS - Simon Williamson Clinic, PC - Birmingham Site Number : 8400004, Birmingham, Alabama
  - Optimal Research Alabama Site Number : 8400019, Huntsville, Alabama
  - Peninsula Research Associates, Inc. Site Number : 8400021, Rolling Hills Estates, California
  - Synexus Clinical Research US, Inc. Site Number : 8400013, Centennial, Colorado
  - Optimal Research, LLC Site Number : 8400002, Melbourne, Florida
  - Synexus Clinical Research US, Inc. - Orlando Site Number : 8400020, Orlando, Florida
  - AES St. Petersburg Site Number : 8400017, Pinellas Park, Florida
  - Synexus Clinical Research US, Inc. - Atlanta Site Number : 8400005, Atlanta, Georgia
  - Synexus Clinical Research Chicago Site Number : 8400012, Chicago, Illinois
  - Synexus Clinical Research Evansville Site Number : 8400008, Evansville, Indiana
  - Synexus St. Louis Site Number : 8400006, St Louis, Missouri
  - Synexus Clinical Research US, Inc. - Henderson Site Number : 8400018, Henderson, Nevada
  - Rochester Clinical Research, Inc. Site Number : 8400023, Rochester, New York
  - Synexus Akron Site Number : 8400009, Akron, Ohio
  - Synexus Clinical Research US, Inc. - Cincinnati Site Number : 8400010, Cincinnati, Ohio
  - Synexus US Columbus Site Number : 8400011, Columbus, Ohio
  - Synexus Clinical Research Anderson Site Number : 8400007, Anderson, South Carolina
  - Coastal Carolina Research Center - N Charleston Site Number : 8400022, North Charleston, South Carolina
  - American Indian Clinical Trials Research Network Site Number : 8400025, Rapid City, South Dakota
  - AES Austin Site Number : 8400003, Austin, Texas
  - Synexus Dallas Site Number : 8400014, Dallas, Texas
  - Synexus Clinical Research US, Inc. - San Antonio Site Number : 8400015, San Antonio, Texas
  - AES Salt Lake City Site Number : 8400016, Murray, Utah
- Colombia (11):
  - Investigational Site Number : 1700010, Aguazul
  - Investigational Site Number : 1700002, Barranquilla
  - Investigational Site Number : 1700008, Barranquilla
  - Investigational Site Number : 1700001, Bogotá
  - Investigational Site Number : 1700005, Cali
  - Investigational Site Number : 1700006, Chía
  - Investigational Site Number : 1700004, Floridablanca
  - Investigational Site Number : 1700007, Girardot
  - Investigational Site Number : 1700009, Meta
  - Investigational Site Number : 1700015, Quindío
  - Investigational Site Number : 1700003, Soledad
- Ghana (3):
  - Investigational Site Number : 2880002, Kintampo
  - Investigational Site Number : 2880003, Kumasi
  - Investigational Site Number : 2880001, Navrongo
- Honduras (2):
  - Investigational Site Number : 3400001, Municipio Del Distrito Central
  - Investigational Site Number : 3400002, San Pedro Sula
- India (10):
  - Investigational Site Number : 3560010, Ajmer
  - Investigational Site Number : 3560002, Ambawadi
  - Investigational Site Number : 3560007, Belagavi
  - Investigational Site Number : 3560001, Jaipur
  - Investigational Site Number : 3560005, Kanpur
  - Investigational Site Number : 3560009, Nagpur
  - Investigational Site Number : 3560011, Odisha
  - Investigational Site Number : 3560004, Patna
  - Investigational Site Number : 3560003, Punjagutta
  - Investigational Site Number : 3560006, Tamilnadu
- Japan (5):
  - Investigational Site Number : 3920005, Chiyoda-ku,, Tokyo
  - Investigational Site Number : 3920004, Haramachi,Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920003, Kouenji minami,Suginami-ku, Tokyo
  - Investigational Site Number : 3920001, Kyobashi Chuo-ku, Tokyo
  - Investigational Site Number : 3920002, Ohta-ku, Tokyo
- Kenya (10):
  - Investigational Site Number : 4040011, Butere
  - Investigational Site Number : 4040006, Eldoret
  - Investigational Site Number : 4040004, Kericho
  - Investigational Site Number : 4040002, Kisumu
  - Investigational Site Number : 4040003, Kisumu
  - Investigational Site Number : 4040012, Kisumu
  - Investigational Site Number : 4040008, Mombasa
  - Investigational Site Number : 4040001, Nairobi
  - Investigational Site Number : 4040007, Nairobi
  - Investigational Site Number : 4040009, Thika
- Mexico (7):
  - Investigational Site Number : 4840005, León, Guanajuato
  - Investigational Site Number : 4840004, Acapulco de Juárez, Guerrero
  - Investigational Site Number : 4840003, Guadalajara, Jalisco
  - Investigational Site Number : 4840009, Mexico City, Mexico City
  - Investigational Site Number : 4840008, Cuernavaca, Morelos
  - Investigational Site Number : 4840006, Temixco
  - Investigational Site Number : 4840002, Veracruz
- Nepal (3):
  - Investigational Site Number : 5240002, Dhulikhel
  - Investigational Site Number : 5240003, Kathmandu
  - Investigational Site Number : 5240001, Nepalgunj
- Uganda (8):
  - Investigational Site Number : 8000002, Entebbe
  - Investigational Site Number : 8000005, Entebbe
  - Investigational Site Number : 8000001, Kampala
  - Investigational Site Number : 8000013, Kampala
  - Investigational Site Number : 8000007, Kampala
  - Investigational Site Number : 8000003, Kampala
  - Investigational Site Number : 8000004, Kampala
  - Investigational Site Number : 8000014, Lira
- Ukraine (4):
  - Investigational Site Number : 8040002, Kiev
  - Investigational Site Number : 8040004, Kyiv
  - Investigational Site Number : 8040003, Kyiv
  - Investigational Site Number : 8040001, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dayan GH, Rouphael N, Walsh SR, Chen A, Grunenberg N, Allen M, Antony J, Asante KP, Bhate AS, Beresnev T, Bonaparte MI, Celle M, Ceregido MA, Corey L, Dobrianskyi D, Fu B, Grillet MH, Keshtkar-Jahromi M, Juraska M, Kee JJ, Kibuuka H, Koutsoukos M, Masotti R, Michael NL, Neuzil KM, Reynales H, Robb ML, Villagomez Martinez SM, Sawe F, Schuerman L, Tong T, Treanor J, Wartel TA, Diazgranados CA, Chicz RM, Gurunathan S, Savarino S, Sridhar S; VAT00008 Study Team. Efficacy of a bivalent (D614 + B.1.351) SARS-CoV-2 recombinant protein vaccine with AS03 adjuvant in adults: a phase 3, parallel, randomised, modified double-blind, placebo-controlled trial. Lancet Respir Med. 2023 Nov;11(11):975-990. doi: 10.1016/S2213-2600(23)00263-1. Epub 2023 Sep 13. PMID 37716365